CLINICAL TRIAL: NCT02494271
Title: TIVA, Inhalation Anesthesia, and Surgical Site Infection
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Dr, Seoul National University Bundang Hospital
Other Study IDs: SSI_anesthesia
Record Dates: First submitted 2015-06-17; First posted 2015-07-10 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-07

CONDITIONS: Colorectal Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Total intravenous anesthesia: Total intravenous anesthesia using propofol and remifentanil
- Inhalation: Balanced inhalation anesthesia using volatile anesthetics and remifentanil

SUMMARY:
The purpose of this retrospective study was to evaluate the incidence of SSI after colorectal surgery under the general anesthesia by different general anesthetic technique: inhalation versus total intravenous anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who underwent elective colorectal surgery under general anesthesia from January 2011 to December 2013.

Exclusion Criteria:

* None

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who underwent elective colorectal surgery under general anesthesia from January 2011 to December 2013 at SNUBH.
Sampling Method: Non-Probability Sample
Enrollment: 2046 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Surgical site infection | Postoperative 30 day
  Number of participants with surgical site infection

SECONDARY OUTCOMES:
Postoperative C-reactive protein | Postoperative 1 day
  Plasma concentration
Segmented neutrophil count | Preoperaitve 1 day, postoperative 1 day
  Segmented neutrophil count
Transfusion | The day of operation, postoperative 30 day
  Number of unit of transfused red blood cells

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea